CLINICAL TRIAL: NCT03441269
Title: A Prospective Randomized Double-Blind Trial Comparing 3 Doses of Oral Ibuprofen in Management of Mild to Moderate Pain in Adult Patients in the ED
Brief Title: Adult Oral Ibuprofen Study for ED Pain Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Antonios Likourezos (Other)
Responsible Party: Sponsor-Investigator, Antonios Likourezos, Research Manager, Maimonides Medical Center
Organization: Maimonides Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-08-04
Record Dates: First submitted 2018-02-15; First posted 2018-02-22 (Actual); Results first posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Pain, Acute
Keywords: Emergency Medicine; Acute Pain; Oral Ibuprofen
MeSH Terms: conditions — Acute Pain | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- 400mg/dose (Active Comparator): Oral Ibuprofen dose of 400mg/dose for mild to moderate acute pain in ED patients.
  Interventions: Drug: Oral Ibuprofen
- 600mg/dose (Active Comparator): Oral Ibuprofen dose of 600mg/dose for mild to moderate acute pain in ED patients.
  Interventions: Drug: Oral Ibuprofen
- 800mg/dose (Active Comparator): Oral Ibuprofen dose of 800mg/dose for mild to moderate acute pain in ED patients.
  Interventions: Drug: Oral Ibuprofen

INTERVENTIONS:
Drug: Oral Ibuprofen — Oral Ibuprofen will be given to all the arms; only the dosage will be different: 400mg vs. 600mg vs. 800mg

SUMMARY:
Ibuprofen is one of the most widely used non-steroidal anti-inflammatory drug (NSAID) for management of mild -to moderate pain in the ED (acute musculo-skeletal pain, headache, dental pain). Ibuprofen as a representative of NSAID's as a class follows the analgesic ceiling concept that postulates that there is a dose of a drug beyond which any further dosage increase results in no additional analgesic effect. Despite this fact, Ibuprofen may commonly be used at doses above its analgesic ceiling, although this may not offer an incremental analgesic advantage and potentially adds risk of harm. The analgesic ceiling dose for ibuprofen is only 200-400mg/dose, and about 1200 mg/day. Thus, we hypothesize that administration of Ibuprofen in a dose of 400 mg in the ED is as effective in treating mild-to-moderate acute pain in patients presenting to the ED as 600 mg and 800 mg

DETAILED DESCRIPTION:
STUDY DESIGN A randomized, double-blind trial to determine the analgesic equivalency of orally administered ibuprofen at 400 mg for the treatment of acute pain in comparison to with higher doses of 600 and 800 mg for managing mild-to-moderate pain of adult patients in the ED.

OUTCOME MEASURES The primary outcome will be reduction in numeric rating scale pain score at 60 minutes from medication administration. Secondary outcomes included rates and percentages of subjects experiencing adverse effects as well as percentage of patients requiring rescue analgesia

STUDY POPULATION Patients considered for inclusion will comprise adults aged 18 and older years who presented to the ED primarily for management of acute mild to moderate musculoskeletal pain, headache, or dental pain who would routinely be treated with oral iburpofen in our ED as determined by the treating attending or resident physician. Acute pain will be defined in our study as having an onset within 30 days or less. Exclusion criteria will include pregnancy or breastfeeding, active peptic ulcer disease, acute gastrointestinal hemorrhage, known history of severe renal or hepatic insufficiency, allergy to nonsteroidal anti-inflammatory drugs, and patients having already received analgesic medication. For the purposes of this study, ibuprofen will be used without co-administration of any other analgesics, with the exception of rescue medication.

STUDY LOCATION The study will be conducted at a 711-bed urban community teaching hospital with an annual ED census of greater than 120,000 visits.

DURATION OF ENROLLMENT Patients pain scores will be recorded at the beginning of the study and at 60 minutes post-administration of medication by utilizing NRS.

DESCRIPTION OF INTERVENTION AND ADMINISTRATION Once the patient is triaged, an initial pain score will be assessed. Patients will then have an initial evaluation by ED physician and, once deemed eligible for the study, the patient will be randomized to receive oral ibuprofen at a dose of 400mg, 600mg, or 800mg. The on-duty ED pharmacist will prepare 400 mg, 600 mg and 800 mg oral ibuprofen preparations in identical capsules according to predetermined randomization generated in SPSS by the research manager. Demographics, chief complaint and initial pain score will be recorded in the data sheet as well as prior analgesics use. Patients pain scores will be recorded at the beginning of the study and at 60 minutes post-administration by using NRS.

RANDOMIZATION/BLINDING The research manager and statistician independently of data collection will conduct the programming of the randomization list, confirmation of written consent acquisition, and statistical analyses. ED pharmacy investigators will maintain the randomization list, prepare the medication, and deliver it to the nurse caring for the study participant in a blinded manner. The preparing pharmacist, research manager, and statistician will be the only ones with knowledge of the study arm to which the participant would be randomized. Providers, participants, and the data-collecting research team will be blinded to the medication received. Study investigators will include treating physicians who will assisted in screening and supervising the research fellow, residents, and research coordinators, who will enroll patients and record pain scores and adverse effects at baseline and at 60 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Adult ED patients aged 18 and older
* Chief complaint of mild to moderate musculoskeletal pain, headache, or dental pain intensity of less than 4 on a standard 0 to 10 numeric rating scale.
* Acute pain (within 30 days of onset)
* Patients who would routinely be treated with oral ibuprofen

Exclusion Criteria:

* pregnancy or breastfeeding,
* active peptic ulcer disease,
* acute gastrointestinal hemorrhage,
* known history of severe renal or hepatic insufficiency, allergy to nonsteroidal anti-inflammatory drugs,
* patients having already received analgesic medication.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Motov, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Motov S, Masoudi A, Drapkin J, Sotomayor C, Kim S, Butt M, Likourezos A, Fassassi C, Hossain R, Brady J, Rothberger N, Flom P, Marshall J. Comparison of Oral Ibuprofen at Three Single-Dose Regimens for Treating Acute Pain in the Emergency Department: A Randomized Controlled Trial. Ann Emerg Med. 2019 Oct;74(4):530-537. doi: 10.1016/j.annemergmed.2019.05.037. Epub 2019 Aug 2. PMID 31383385

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 400mg/Dose | 600mg/Dose | 800mg/Dose
Started | 75 | 75 | 75
Completed | 75 | 74 | 74
Not Completed | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 400mg/Dose | 600mg/Dose | 800mg/Dose | Total
Number analyzed (Participants) | 75 | 75 | 75 | 225
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.9 (16.2) | 45.6 (15.8) | 42.6 (15.9) | 44.4 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 44 | 28 | 111
  Male | 36 | 31 | 47 | 114
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 75 | 75 | 75 | 225

OUTCOME MEASURES:

1. Primary Outcome: Pain Reduction at 60 Minutes From Baseline of the 3 Oral Ibuprofen Groups
Description: Difference in mean pain scores among all groups from at 60 minutes from baseline; negative difference infers decrease in pain score. A pain score of 10 indicates severe pain, 5 indicates moderate pain and 0 indicates no pain.
Time Frame: 60 minutes
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 400mg/Dose | 600mg/Dose | 800mg/Dose
Number analyzed (Participants) | 75 | 74 | 74
units on a scale | -2.12 [-2.45 to -1.80] | -1.85 [-2.05 to -1.66] | -1.96 [-2.18 to -1.74]

2. Secondary Outcome: Rates of Adverse Event of the 3 Oral Ibuprofen Dosage Groups
Description: Rates of Adverse Event of the 3 Oral Ibuprofen Dosage Groups
Time Frame: 60 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | 400mg/Dose | 600mg/Dose | 800mg/Dose
Number analyzed (Participants) | 75 | 74 | 74
Participants | 0 | 0 | 0

3. Secondary Outcome: Rates of Requiring Rescue Analgesia
Description: Rates of Requiring Rescue Analgesia for pain management
Time Frame: 60 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | 400mg/Dose | 600mg/Dose | 800mg/Dose
Number analyzed (Participants) | 75 | 74 | 74
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 60 minutes
Description: Any serious adverse events within 60 minutes after baseline
Arm/Group | 400mg/Dose | 600mg/Dose | 800mg/Dose
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/74 | 0/74
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/74 | 0/74
Other Adverse Events (participants affected / at risk) | 0/75 | 0/74 | 0/74

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/69/NCT03441269/Prot_SAP_000.pdf